CLINICAL TRIAL: NCT03351595
Title: Evaluation of Influencing Factors Affecting Childhood Metabolic Indicators in Korea (Repeated Measures Analysis; Longitudinal Birth Study)
Brief Title: Ewha Birth and Growth Study (Birth Cohort)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ewha Womans University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Other Study IDs: EWCS
Record Dates: First submitted 2017-10-18; First posted 2017-11-24 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Pediatric Health
Keywords: Growth pattern; Environmental and prenatal exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ongoing longitudinal birth cohort established at Mok-dong Hospital, Ewha Woman's University, Seoul, South Korea, between 2001 and 2006.

DETAILED DESCRIPTION:
Cohort composed of mothers, who visited to prenatal care between 24 and 28 weeks of gestation, between 2001 and 2006. After the child was born then, we collected information at birth outcome and conducted mail surveys at 6, 12, 18, and 24 months. Regular check-up was conducted at 3, 5, and every year after 7 years of age(last check up point: 15 years old). In check-up survey, after an 8-hour overnight fast, blood and urine samples (3 ml EDTA-blood and 5 ml serum) were obtained from subjects by venepuncture. following parameters were checked: physical growth, blood pressure. metabolic biomarker(Total cholesterol, HDl-cholesterol, TG(triglyceride), glucose, uric acid, etc.), K-CBCL(Korea-child behavior checklist), 24 hour recall method for nutrition, FFQ(Food Frequency Questionnaire), Questionnaires including Socio-economic status and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Participants' mothers, who visited to prenatal care between 24 and 28 weeks of gestation.
* An individual who can be followed up during the study period and is capable of complying with the study requirements

Exclusion Criteria:

* An individual thought to have difficulty participating in the study due to other reasons, based on the judgment of the investigator

Ages: 24 Weeks to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants and Participants' mothers
Sampling Method: Non-Probability Sample
Enrollment: 734 (Actual)
Dates: Start 2001-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Profile of participants received regular medical check-up and result feed back for growth development | 365days
  Changes from baseline in physical growth using anthropometric measurement

SECONDARY OUTCOMES:
Profile of participants received blood pressure measurement for pediatric hypertension | 365days
  Changes from baseline in average blood pressure(mmHg, diastolic and systolic) as above the 95th percentile adjusted for sex, age, and height percentile

IPD SHARING:
Plan to Share IPD: Undecided